CLINICAL TRIAL: NCT03803540
Title: Fecal Microbiota Transplantation for the Treatment of Non-Alcoholic Steatohepatitis, a Pilot Study.
Brief Title: Fecal Microbiota Transplantation for the Treatment of Non-Alcoholic Steatohepatitis
Acronym: FMT-NASH
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Hospital Universitario Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Jose Luis Calleja, Head of the department of Gastroenterology and Hepatology, Puerta de Hierro University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT-NASH
Record Dates: First submitted 2019-01-09; First posted 2019-01-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non Alcoholic Steatohepatitis
Keywords: Non-Alcoholic Fatty Liver Disease; Non Alcoholic Steatohepatitis; NAFLD; NASH; Fecal Microbiota Transplantation; FMT
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): Lean healthy donor frozen fecal microbiota will be administered via duodenal infusion in an upper gastrointestinal endoscopy
  Interventions: Other: Fecal Microbiota Transplantation

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation via duodenal infusion

SUMMARY:
Human microbiota is the set of microorganisms that, in a symbiotic way, coexist and develop in the different surfaces (skin and mucous membranes) of the human body. It is estimated that it is composed of approximately 10^14 bacteria and other unicellular life forms . The gastrointestinal (GI) tract is the organ in which the microbiota reaches its greatest complexity, influencing its metabolic activities in different organs and human systems.

Human microbiota plays a role in multiple homeostatic and physiological functions including energy and intermediary metabolism, normal immune responses, and even appropriate bowel development and nervous system functioning. Given its vascular supply, the liver plays important roles in metabolism and immunological functions. It receives 70% of blood supply through the portal vein which carries all metabolic products derived from GI microbiota.

Non alcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease in developed countries (with an estimated prevalence around 25 - 40% of adults) and it is expected that the burden of disease will increase in the near future. This condition can progress through a spectrum of progressive liver damage to non alcoholic steatohepatitis (NASH), liver fibrosis, cirrhosis and liver cancer. Around 20-30% of NAFLD patients develop NASH, with a lower rate progressing further to fibrosis and cirrhosis. Currently, there is no approved pharmacological or interventional treatment for the management of this so prevalent disease, apart from changes in lifestyle aiming weight loss.

The aim of the present pilot study is to assess the efficacy and safety of microbiota manipulation by means of Fecal Microbiota Transplantation in the treatment of patients with NASH.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index > 30 Kg / m^2
* Histological evidence of NASH (by means of hepatic percutaneous biopsy obtained in the previous six months) defined as at least 1 point in each category of NAFLD Activity Score with a fibrosis stage between 0 and 3.
* Global NAFLD Activity Score >= 4 points
* For patients with fibrosis stage 0 or 1, NAFLD Activity Score should be >= 5 points and they should have one of the following comorbidities: Metabolic Syndrome, type 2 diabetes mellitus or Homeostasis Model Assessment - Insulin Resistance (HOMA-IR) > 6.

Exclusion Criteria:

* Patients unable or unwilling to give the informed consent
* Patients actively participating in another clinical trial or investigational protocol
* Cirrhosis of the liver: Transient elastography > 20 kilopascal or histological evidence of it (grade 4 fibrosis)
* Alcoholic consumption greater than 14 g / week in women or 21 g / week in men
* Any significant hepatic comorbidity: chronic active viral hepatitis, cholestatic disease, hemochromatosis or Wilson disease
* HIV infection
* Liver transplantation
* Hepatocellular carcinoma
* Women during pregnancy or breastfeeding
* Portal thrombosis
* Non-cirrhotic portal hypertension
* Gastroesophageal varices
* Previous gastrointestinal tract major surgery (excluding appendectomy and cholecystectomy)
* Previous Fecal Microbiota Transplantation
* Chronic significant kidney or heart disease
* Life expectancy lower than two years
* Chronic use of steatogenic drugs
* Chronic use of immunosuppressants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy (Histological resolution of NASH defined as ballooning disappearance with or without persistence of minimal lobulillar inflammation and no progression of fibrosis stage) | 72 weeks
  Two liver biopsy samples (one pre-FMT and the second 72 weeks after FMT) will be taken. Resolution of NASH is defined as ballooning disappearance with or without persistence of minimal lobulillar inflammation and no progression of fibrosis stage. NAFLD Activity Score is the histological scale that will be used.

SECONDARY OUTCOMES:
Safety (Appearance of adverse events related with Fecal Microbiota Transplantation) | 72 weeks
  Appearance of adverse events related with Fecal Microbiota Transplantation will be recorded during 72 weeks follow-up.
Microbiota composition (Changes in microbiota diversity profile related with Fecal Microbiota Transplantation via 16S rRNA analysis) | 72 weeks
  Changes in microbiota diversity profile related with Fecal Microbiota Transplantation procedure. 16S rRNA sequencing techniques will be applied on stool samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Puerta de Hierro University Hospital, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No